CLINICAL TRIAL: NCT02874963
Title: Impact of Combined Non-surgical and Surgical Periodontal Treatment in Patients With Type 2 Diabetes Mellitus
Brief Title: FM-SRP and Tooth Extraction Improve Type 2 Diabetes Mellitus in Periodontitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Clinical Centre of Kosova (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Dashor Bukleta, Oral Surgery Specialist (PhD Candidate), University Clinical Centre of Kosova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUCSK
Record Dates: First submitted 2016-08-01; First posted 2016-08-22 (Estimated); Last update posted 2016-08-22 (Estimated); Status verified 2016-08

CONDITIONS: Periodontitis; Type 2 Diabetes Mellitus
Keywords: Diabetes; Oral Hygiene; Periodontal Surgery; Periodontal Medicine
MeSH Terms: conditions — Periodontitis; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Tooth Extraction; Listerine; Ethanol; methyl salicylate; Menthol; Thymol; Mouthwashes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical periodontal treatment (Active Comparator): Type 2 Diabetes Patients with periodontitis (without initial non-surgical periodontal therapy) at least one tooth extraction will be performed.
  Non-Diabetes Patients with periodontitis (without initial non-surgical periodontal therapy) at least one tooth extraction will be performed.
  Intervention:
  Procedure: Surgery (Tooth Extraction)
  Interventions: Procedure: Surgical Periodontal Treatment
- Surgical and non-surgical periodontal treatment (Active Comparator): Type 2 Diabetes Patients with periodontitis (with initial non-surgical periodontal therapy) at least one tooth extraction will be performed.
  Non-Diabetes Patients with periodontitis (with initial non-surgical periodontal therapy) at least one tooth extraction will be performed.
  Interventions:
  Procedure: Surgery (Tooth Extraction)
  Procedure: Non-surgical periodontal therapy-full mouth scaling and root planing (FM-SRP) with ultrasonic device and periodontal curets for mechanical debridement of the supra- and sub-gingival plaque and calculus, post operative rinsing thrice a day for 3 weeks.
  Interventions: Procedure: Surgical Periodontal Treatment; Device: Non Surgical Periodontal Treatment includes scaling root planing with UDS-J Ultrasonic Scaler.; Drug: Non Surgical Periodontal Treatment includes post operative mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%)

INTERVENTIONS:
Procedure: Surgical Periodontal Treatment — In the patient's with periodontal disease at least one tooth extraction will be performed.
  Other Names: Tooth Extraction
Device: Non Surgical Periodontal Treatment includes scaling root planing with UDS-J Ultrasonic Scaler. — Previous to surgery procedures, in particular in the two groups with an adjunctive non surgical periodontal treatment such as full mouth tooth cleaning will be included: full-mouth scaling and root planing (FM-SRP) with ultrasonic device (UDS-J Ultrasonic Scaler, Guilin Woodpecker Medical Instrument) and periodontal curets for mechanical debridement of the supra- and sub-gingival plaque and calculus.
  Other Names: FM-SRP
  Arms: Surgical and non-surgical periodontal treatment
Drug: Non Surgical Periodontal Treatment includes post operative mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%) — Previous to surgery procedures, in particular in the two groups with an adjunctive non surgical periodontal treatment such as full mouth tooth cleaning will be included mouth wash with Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%) for the 3 weeks after tooth extraction and cleaning.
  Other Names: Mouth wash
  Arms: Surgical and non-surgical periodontal treatment

SUMMARY:
This intervention study is designed to evaluate the effects of non-surgical procedure in addition to surgical procedure on systemic inflammation and glycemic control in with type 2 diabetes mellitus patients with periodontitis in comparison with non-diabetic periodontic patients.

DETAILED DESCRIPTION:
In a randomize, prospective study 200 patients from the endocrinology department of "Peja's Regional Hospital" and Dental Polyclinic at city of Peja, will be assessed and examined for eligibility. Personal interviews will be used to collect the baseline data from each participant using a pre structured questionnaire.

After clinical examination, 160 patients aged 30-70 years will be selected for the study. These will be further divided in four groups: type 2 diabetes mellitus group (with or without initial periodontal therapy) and non-diabetic group (with or without initial periodontal therapy).

All the patients will be with periodontal disease and at least one tooth extraction will perform. Previous to surgery procedures, in particular in the two groups with an adjunctive non surgical periodontal treatment such as full mouth tooth cleaning will be included: full-mouth scaling and root planing (FM-SRP) with ultrasonic device (UDS-J Ultrasonic Scaler, Guilin Woodpecker Medical Instrument) and periodontal curets for mechanical debridement of the supra- and sub-gingival plaque and calculus.

Post operative rinsing will be followed with antiseptic solution Listerine® (ethanol 21.6%, methyl salicylate 0.06%, menthol 0.042%, thymol 0.064% and eucalyptol 0.092%) as a mouthwash thrice a day for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 Diabetes Mellitus; having a baseline HbA1c ≥ 6.5%, at least 10 teeth in the functional dentition (excluding third molars) and a clinical diagnosis of periodontal disease with at least one site with probing depth (PD) ≥ 5mm, and two teeth with attachment lost ≥ 6mm and no modification in the pharmacological treatment of diabetes during the study period.

Exclusion Criteria:

* Pregnancy or lactation, major diabetic complications, uses of antibiotic therapy or non-steroidal anti-inflammatory drug therapy 4 months before the first visit.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2015-11; Primary Completion 2016-09 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Biochemical parameter: HbA1c (mean value in %), | Baseline and 3 months after
  The changes in levels of glycated haemoglobin after periodontal treatment.
Biochemical parameter: high sensitive C-Reactive Protein - hs-CRP (mean value in mg/L) | Baseline and 3 months after
  The changes in levels of c-reactive protein after periodontal treatment.

SECONDARY OUTCOMES:
Bleeding on probing (BOP) (expressed in %) | Baseline and 3 months after
  The changes in bleeding on probing after periodontal treatment.
Mean attachment level (MAL) (mean in mm, as a measure of periodontal parameter) | Baseline and 3 months after
  The changes in clinical attachment level after periodontal treatment.
Plaque index (PI) (expressed in %) | Baseline and 3 months after
  The changes in plaque index after periodontal treatment.
Mean probing depth (PD) (mean in mm, as a measure of periodontal parameter) | Baseline and 3 months after
  The changes in probing pocket depth after periodontal treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Dashnor Bukleta, Dr, Principal Investigator — Department of Oral Medicine and Periodontology, Faculty of Medicine, University of Ljubljana, Ljubljana, Slovenia
Locations (1):
- Oral Surgery, Dental Polyclinic (HUCSK), Peja, Kosovo

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] American Diabetes Association. Executive summary: Standards of medical care in diabetes--2014. Diabetes Care. 2014 Jan;37 Suppl 1:S5-13. doi: 10.2337/dc14-S005. No abstract available. PMID 24357214
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Zeqiri S, Ylli A, Zeqiri N. The effect of physical activity in glycemia in patients with diabetes mellitus. Med Arh. 2007;61(3):146-9. PMID 18232276
- [Background] Jerliu N, Toci E, Burazeri G, Ramadani N, Brand H. Prevalence and socioeconomic correlates of chronic morbidity among elderly people in Kosovo: a population-based survey. BMC Geriatr. 2013 Mar 1;13:22. doi: 10.1186/1471-2318-13-22. PMID 23452830
- [Background] Daci A, Elshani B, Giangiacomo B. Gestational diabetes mellitus (GDM) in the Republic of Kosovo: a retrospective pilot study. Med Arch. 2013;67(2):88-90. doi: 10.5455/medarh.2013.67.88-90. PMID 24341050
- [Background] Albert DA, Ward A, Allweiss P, Graves DT, Knowler WC, Kunzel C, Leibel RL, Novak KF, Oates TW, Papapanou PN, Schmidt AM, Taylor GW, Lamster IB, Lalla E. Diabetes and oral disease: implications for health professionals. Ann N Y Acad Sci. 2012 May;1255:1-15. doi: 10.1111/j.1749-6632.2011.06460.x. Epub 2012 Mar 12. PMID 22409777
- [Background] Mealey BL, Oates TW; American Academy of Periodontology. Diabetes mellitus and periodontal diseases. J Periodontol. 2006 Aug;77(8):1289-303. doi: 10.1902/jop.2006.050459. PMID 16881798
- [Background] Loe H. Periodontal disease. The sixth complication of diabetes mellitus. Diabetes Care. 1993 Jan;16(1):329-34. No abstract available. PMID 8422804
- [Background] Tsai C, Hayes C, Taylor GW. Glycemic control of type 2 diabetes and severe periodontal disease in the US adult population. Community Dent Oral Epidemiol. 2002 Jun;30(3):182-92. doi: 10.1034/j.1600-0528.2002.300304.x. PMID 12000341
- [Background] Touger-Decker R, Schaefer M, Flinton R, Steinberg L. Effect of tooth loss and dentures On diet habits. J Prosthet Dent 1996;75:831.
- [Background] Kamberi B, Hoxha V, Stavileci M, Dragusha E, Kuci A, Kqiku L. Prevalence of apical periodontitis and endodontic treatment in a Kosovar adult population. BMC Oral Health. 2011 Nov 29;11:32. doi: 10.1186/1472-6831-11-32. PMID 22126237
- [Background] Begzati A, Meqa K, Siegenthaler D, Berisha M, Mautsch W. Dental health evaluation of children in kosovo. Eur J Dent. 2011 Jan;5(1):32-9. PMID 21228954
- [Background] Saremi A, Nelson RG, Tulloch-Reid M, Hanson RL, Sievers ML, Taylor GW, Shlossman M, Bennett PH, Genco R, Knowler WC. Periodontal disease and mortality in type 2 diabetes. Diabetes Care. 2005 Jan;28(1):27-32. doi: 10.2337/diacare.28.1.27. PMID 15616229
- [Background] Pucher J, Stewart J. Periodontal disease and diabetes mellitus. Curr Diab Rep. 2004 Feb;4(1):46-50. doi: 10.1007/s11892-004-0011-y. PMID 14764280
- [Background] Norris SL, Engelgau MM, Narayan KM. Effectiveness of self-management training in type 2 diabetes: a systematic review of randomized controlled trials. Diabetes Care. 2001 Mar;24(3):561-87. doi: 10.2337/diacare.24.3.561. PMID 11289485
- [Background] Soskolne WA, Klinger A. The relationship between periodontal diseases and diabetes: an overview. Ann Periodontol. 2001 Dec;6(1):91-8. doi: 10.1902/annals.2001.6.1.91. PMID 11887477
- [Background] Khader YS, Al Habashneh R, Al Malalheh M, Bataineh A. The effect of full-mouth tooth extraction on glycemic control among patients with type 2 diabetes requiring extraction of all remaining teeth: a randomized clinical trial. J Periodontal Res. 2010 Dec;45(6):741-7. doi: 10.1111/j.1600-0765.2010.01294.x. PMID 20682017
- [Background] Nesto R. C-reactive protein, its role in inflammation, Type 2 diabetes and cardiovascular disease, and the effects of insulin-sensitizing treatment with thiazolidinediones. Diabet Med. 2004 Aug;21(8):810-7. doi: 10.1111/j.1464-5491.2004.01296.x. PMID 15270782
- [Background] Paraskevas S, Huizinga JD, Loos BG. A systematic review and meta-analyses on C-reactive protein in relation to periodontitis. J Clin Periodontol. 2008 Apr;35(4):277-90. doi: 10.1111/j.1600-051X.2007.01173.x. Epub 2008 Feb 20. PMID 18294231
- [Background] Grossi SG, Genco RJ. Periodontal disease and diabetes mellitus: a two-way relationship. Ann Periodontol. 1998 Jul;3(1):51-61. doi: 10.1902/annals.1998.3.1.51. PMID 9722690
- [Background] Corbella S, Francetti L, Taschieri S, De Siena F, Fabbro MD. Effect of periodontal treatment on glycemic control of patients with diabetes: A systematic review and meta-analysis. J Diabetes Investig. 2013 Sep 13;4(5):502-9. doi: 10.1111/jdi.12088. Epub 2013 Apr 18. PMID 24843701
- [Background] Kiran M, Arpak N, Unsal E, Erdogan MF. The effect of improved periodontal health on metabolic control in type 2 diabetes mellitus. J Clin Periodontol. 2005 Mar;32(3):266-72. doi: 10.1111/j.1600-051X.2005.00658.x. PMID 15766369
- [Background] Teeuw WJ, Gerdes VE, Loos BG. Effect of periodontal treatment on glycemic control of diabetic patients: a systematic review and meta-analysis. Diabetes Care. 2010 Feb;33(2):421-7. doi: 10.2337/dc09-1378. PMID 20103557
- [Background] Wang X, Han X, Guo X, Luo X, Wang D. The effect of periodontal treatment on hemoglobin a1c levels of diabetic patients: a systematic review and meta-analysis. PLoS One. 2014 Sep 25;9(9):e108412. doi: 10.1371/journal.pone.0108412. eCollection 2014. PMID 25255331